CLINICAL TRIAL: NCT02140151
Title: Prophylactic Ranibizumab for Exudative Age-related Macular Degeneration (AMD) in Vulnerable Eyes With Nonexudative AMD Trial: A Multicenter, Prospectively Randomized, Masked and Controlled, Interventional Investigator Sponsored Phase I/II Study
Brief Title: Prophylactic Ranibizumab for Exudative Age-related Macular Degeneration
Acronym: PREVENT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Southern California Desert Retina Consultants, MC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ML29258
Record Dates: First submitted 2014-04-25; First posted 2014-05-16 (Estimated); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Age-related Macular Degeneration
Keywords: amd; non-exudative macular degeneration; exudative macular degeneration; age-related macular degeneration; ranibizumab; anti-VEGF
MeSH Terms: conditions — Macular Degeneration; Glycogen Storage Disease Type II; Wet Macular Degeneration | interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sham (No Intervention): Sham Injection
- Quarterly Ranibizumab 0.5mg (Active Comparator): Quarterly intravitreal injection of 0.5mg ranibizumab
  Interventions: Drug: Ranibizumab 0.5mg

INTERVENTIONS:
Drug: Ranibizumab 0.5mg
  Other Names: Lucentis
  Arms: Quarterly Ranibizumab 0.5mg

SUMMARY:
This study will determine whether quarterly injections of Ranibizumab may prevent eyes with dry age-related macular degeneration from progressing to wet age-related macular degeneration (AMD).

DETAILED DESCRIPTION:
This is a multicenter, prospectively randomized, masked and controlled, interventional investigator sponsored phase I/II study of subjects with high-risk nonexudative age-related macular degeneration (AMD) treated with intravitreal ranibizumab quarterly for prophylaxis of conversion to exudative age-related macular degeneration.

The objective of this study is to investigate the safety and efficacy of prophylactic anti-vascular endothelial growth factor (VEGF) therapy with ranibizumab to prevent the development of exudative AMD in eyes with high-risk nonexudative AMD. In addition, baseline characteristics of high-risk eyes (fundus features, optical coherence tomography (OCT) parameters and genetic profile) will be evaluated to determine their predictive value in conversion to exudative AMD. The effect of ranibizumab on the atrophic component of AMD will also be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Adult over 50 years old
* Able to sign informed consent and comply with the study protocol for the duration of two years
* Nonexudative age-related macular degeneration (AMD) in one eye (study eye)
* History of exudative AMD in one eye only (fellow eye) diagnosed within 5 years of study enrollment

Exclusion Criteria:

* Participation in another simultaneous medical investigation or clinical trial
* Patient is pregnant, lactating, or premenopausal and not using adequate contraception
* Known serious allergies to ranibizumab, fluorescein dye, drugs for pupillary dilation, topical anesthetic, sterilizing solution (e.g. Betadine solution)
* Presence of ocular conditions with increased risk of choroidal neovascularization (CNVM) or pigment epithelial detachment (PED), including presumed ocular histoplasmosis syndrome (POHS), traumatic choroidal rupture, angioid streaks, pathologic myopia (spherical equivalent of ≥ -8 diopters or axial length of ≥ 25 mm), multifocal choroiditis, macular choroidal nevus, polypoidal choroidal vasculopathy (PCV), idiopathic central serous chorioretinopathy (ICSC), etc.
* History of vitrectomy in the study eye
* History of cataract surgery within 3 months of enrollment
* History of yttrium aluminum garnet (YAG) capsulotomy within 1 month of enrollment
* History of intraocular or periocular corticosteroid therapy within the past 90 days
* History of therapeutic radiation in the region of the study eye.
* Presence of media opacity that would preclude adequate examination and/or imaging
* Concurrent macular conditions that would affect the study parameters (epiretinal membrane, macular hole, macular edema) or require treatment within the duration of the study
* Any progressive ocular condition (uncontrolled glaucoma, diabetic retinopathy, uveitis) that may affect the visual acuity for the duration of the study
* Active ocular infection (i.e., bacterial, viral, parasitic, or fungal) in either eye at enrollment
* Presence of any advanced systemic condition that may hinder the patients participation and completion of the study
* Concurrent use of systemic anti-VEGF therapy

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2014-09-17 (Actual); Primary Completion 2020-07-09 (Actual); Study Completion 2020-07-09 (Actual)

PRIMARY OUTCOMES:
Development of exudative AMD | 2 years
  Development of choroidal neovascularization (conversion) defined by the presence of leakage on fluorescein angiography (FA) and fluid within or below the retina or below the retinal pigment epithelium seen on spectral-domain optical coherence tomography (SD-OCT)

SECONDARY OUTCOMES:
Vision change | 2 years
  Change in best-corrected visual acuity (BCVA) from baseline at 12 and 24 months
Vision loss | 2 years
  Proportion of eyes losing < 5, 10, and 15 letters on EDTRS chart at 12 and 24 months
Number of injections | 2 years
  Number of injections required in eyes that convert from dry to wet AMD during the study period
Baseline predictive factors | 2 years
  Baseline demographic, genetic and ocular characteristics predictive of development of wet AMD
Development of geographic atrophy (GA) | 2 years
  Development of geographic atrophy (GA) as detected by fundus photography (FP) and/or fundus autofluorescence (AF).
Ocular adverse events | 2 years
  Incidence and severity of ocular adverse events, as identified by eye examination and imaging
Systemic adverse events | 2 years
  Incidence and severity of other adverse events, as identified by physical examination or subject reporting.

CONTACTS AND LOCATIONS:
Overall Officials: Maziar Lalezary, MD, Principal Investigator — Southern California Desert Retina Consultants
Locations (4):
- United States (4):
  - Northern California Retina Vitreous Associates, Mountain View, California
  - Southern California Desert Retina Consultants, Palm Desert, California
  - Elman Retina, Baltimore, Maryland
  - Black Hills Regional Eye Institute, Rapid City, South Dakota